CLINICAL TRIAL: NCT03975595
Title: Meditation Effects on Brain Function in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Maryland, Baltimore (Other); University of California, San Diego (Other); University of Utah (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB00192687; R61AT010134 (NIH)
Record Dates: First submitted 2019-05-30; First posted 2019-06-05 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation Group A (Active Comparator): A brief meditation intervention involving guided breathing and/or attention exercises (further information withheld to preserve blinding).
  Meditation Group A is the Savoring Meditation Condition. Participants in this condition were trained to generate positive emotions through savoring a pleasant autobiographical memory in a multi-sensory manner.
  Interventions: Behavioral: Meditation Intervention A
- Meditation Group B (Active Comparator): A brief meditation intervention involving guided breathing and/or attention exercises (further information withheld to preserve blinding).
  Meditation Group B is the Breathing Meditation Condition. Participants in this condition were trained to relax and body and take deep breaths in a self-directed manner.
  Interventions: Behavioral: Meditation Intervention B

INTERVENTIONS:
Behavioral: Meditation Intervention A — This will be a brief meditation intervention involving guided breathing and/or attention exercises. Further information is withheld to preserve blinding.
  Arms: Meditation Group A
Behavioral: Meditation Intervention B — This will be a brief meditation intervention involving guided breathing and/or attention exercises. Further information is withheld to preserve blinding.
  Arms: Meditation Group B

SUMMARY:
The purpose of this study is to determine the neural mechanisms supporting meditation-based pain relief in rheumatoid arthritis (RA) patients. The scientific premise is that RA patients' use of different meditation practices during noxious thermal stimulation will alter neural function in brain areas associated with pain, evaluation, and emotional appraisal. The investigators will randomize RA patients to a brief 4-session course of Intervention A (n=20) or Intervention B (n=20). At post-intervention, participants will undergo functional MRI (fMRI) using a perfusion-based arterial spin labeling (ASL) technique during noxious thermal stimulation to determine if the meditation practices differentially alter neural function during noxious thermal stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Withheld to preserve recruitment integrity.

Exclusion Criteria:

* Withheld to preserve recruitment integrity.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Campbell, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Meditation Group A-Savoring: A brief meditation intervention involving guided breathing and/or attention exercises (further information withheld to preserve blinding).
  Meditation Intervention A: This will be a brief meditation intervention involving guided breathing and/or attention exercises. Further information is withheld to preserve blinding.
  Participants in the Savoring Meditation Condition were trained to generate positive emotions through savoring a positive autobiographical memory in a multi-sensory manner.
- Meditation Group B-Breathing: A brief meditation intervention involving guided breathing and/or attention exercises (further information withheld to preserve blinding).
  Meditation Intervention B: This will be a brief meditation intervention involving guided breathing and/or attention exercises. Further information is withheld to preserve blinding.
  Participants in the Breathing Meditation condition were trained to relax the body and take deep breaths in a self-directed manner.
Period: Overall Study
Arm/Group | Meditation Group A-Savoring | Meditation Group B-Breathing
Started | 21 | 23
Completed | 15 | 14
Not Completed | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Meditation Group A: A brief meditation intervention involving guided breathing and/or attention exercises (further information withheld to preserve blinding).
  Meditation Group A is the Savoring Meditation Condition. Participants in this condition were trained to generate positive emotions through savoring a pleasant autobiographical memory in a multi-sensory manner.
  Meditation Intervention A: This will be a brief meditation intervention involving guided breathing and/or attention exercises. Further information is withheld to preserve blinding.
- Meditation Group B: A brief meditation intervention involving guided breathing and/or attention exercises (further information withheld to preserve blinding).
  Meditation Group B is the Breathing Meditation Condition. Participants in this condition were trained to relax and body and take deep breaths in a self-directed manner.
  Meditation Intervention B: This will be a brief meditation intervention involving guided breathing and/or attention exercises. Further information is withheld to preserve blinding.
- Total: Total of all reporting groups
Arm/Group | Meditation Group A | Meditation Group B | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (12.0) | 49.8 (10.9) | 50.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 5 | 5 | 10
  Race: White or European American | 13 | 13 | 26
  Race: Other | 2 | 3 | 5
  Race: Asian | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Lateral Orbital Frontal Cortex Activation
Description: Activation in the Lateral Orbital Frontal Cortex will be quantitatively measured as the difference in cerebral blood flow (CBF) response during noxious thermal stimulation while participants actively practice Intervention A in the scanner, compared to the CBF response during noxious thermal stimulation while participants rest. The unit of measure will be milliliter per 100 gram brain tissue per minute.
Time Frame: Measured at the post-Intervention time point during an MRI scan, approximately 60 minutes.
Population: This outcome was not assessed because it was intended for comparison with a treatment arm (mindful breathing) that was dropped from the study due to COVID-19 delays. No data was collected.
Groups:
- Meditation Group A: A brief meditation intervention involving guided breathing and/or attention exercises (further information withheld to preserve blinding).
  Meditation Intervention A: This will be a brief meditation intervention involving guided breathing and/or attention exercises. Further information is withheld to preserve blinding.
- Meditation Group B: A brief meditation intervention involving guided breathing and/or attention exercises (further information withheld to preserve blinding).
  Meditation Intervention B: This will be a brief meditation intervention involving guided breathing and/or attention exercises. Further information is withheld to preserve blinding.
Arm/Group | Meditation Group A | Meditation Group B
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Nucleus Accumbens Activation
Description: Activation in the Nucleus Accumbens will be quantitatively measured as the difference in cerebral blood flow (CBF) response during noxious thermal stimulation while participants actively practice Intervention B in the scanner, compared to the CBF response during noxious thermal stimulation while participants rest. The unit of measure will be milliliter per 100 gram brain tissue per minute (ml/100g/min). There is no normal range for this measure.
Time Frame: Measured at the post-Intervention time point during an MRI scan, approximately 60 minutes
Measure: Mean (Standard Deviation); unit: ml/100g/min
Arm/Group | Meditation Group A-Savoring | Meditation Group B-Breathing
Number analyzed (Participants) | 15 | 14
ml/100g/min | 16153.59 (1309.90) | 15834.56 (1681.54)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the duration of the study, approximately 4-6 weeks per participant.
Arm/Group | Meditation Group A-Savoring | Meditation Group B-Breathing
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 0/21 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT03975595/Prot_SAP_000.pdf